CLINICAL TRIAL: NCT01573663
Title: Open Label, Randomized, 3-sequence Crossover Study to Evaluate the Drug-drug Interaction Between Ambroxol HCl and Levodropropizine in Healthy Male Volunteers
Brief Title: A Drug-Drug Interaction Study of Ambroxol and Levodropropizine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HM-AMBLE-101
Record Dates: First submitted 2012-04-05; First posted 2012-04-09 (Estimated); Last update posted 2012-07-19 (Estimated); Status verified 2012-04

CONDITIONS: Healthy
Keywords: Ambroxol; Levodropropizine; Drug-drug interaction
MeSH Terms: interventions — Ambroxol; dipropizine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Ambroxol and Levodropropizine (Experimental)
  Interventions: Drug: Ambroxol and Levodropropizine
- Ambroxol (Active Comparator)
  Interventions: Drug: Ambroxol
- Levodropropizine (Active Comparator)
  Interventions: Drug: Levodropropizine

INTERVENTIONS:
Drug: Ambroxol and Levodropropizine — Ambroxol HCl 30mg & Levodropropizine 60mg, PO, Single dose
  Arms: Ambroxol and Levodropropizine
Drug: Ambroxol — Ambroxol HCl 30mg, PO, single dose
  Arms: Ambroxol
Drug: Levodropropizine — Levodropropizine 60mg, PO, single dose
  Arms: Levodropropizine

SUMMARY:
The purpose of this study is to evaluate the drug-durg interaction between ambroxol and levodropropizine.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male
* Age between 20 and 55
* Signed informed consent

Exclusion Criteria:

* Has a history of hypersensitivity to IP ingredients
* Hypotension or hypertension
* Has a history of acute infection within 14 days of screening

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2012-02; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
AUClast | 0-48hrs
Cmax | 0-48hrs

SECONDARY OUTCOMES:
Tmax | 0-48hrs
T1/2 | 0-48hrs
AUCinf | 0-48hrs

CONTACTS AND LOCATIONS:
Overall Officials: Wooseong Huh, MD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung medical center, Seoul, South Korea